CLINICAL TRIAL: NCT03508115
Title: Changes in Cognition in HCV Patients After Virus Eradication With Direct Antiviral Agents. Relationship With Clinical and Sociodemographic Variables
Brief Title: Changes in Cognition in HCV Patients After Virus Eradication With Direct Antiviral Agents
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Mercè Jodar-Vicente, Clinical Neuropsychologist, Corporacion Parc Tauli
Other Study IDs: CIR2015/042
Record Dates: First submitted 2018-03-28; First posted 2018-04-25 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: HCV Infection; HCV Coinfection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Study about the improvement of cognitive, psychopathological and functional abilities in Hepatitis C Virus (HCV) infected patients after eradication of the virus with direct antiviral agents.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect that the eradication of the HCV has on cognition, quality of life and psychopathology. At the same time, investigators intend to study the association between cognitive changes and some clinical variables.

The sample consists of 80 subjects (40 HCV patients and 40 HCV patients coinfected with the Human Immunodeficiency Virus, HIV). Exclusion criteria: Cirrhosis, presence of minimal hepatic encephalopathy or active drug consumption.

A neuropsychological assessment is made before the treatment with direct antiviral agents to evaluate memory, executive functions, processing speed, anxiety, depression and quality of life. Additionally, the following clinical variables are collected: Viral charge, immunosuppression (measured with T Cells CD4 (CD4), CD4 nadir and T Cells CD8 (CD8)) and fibrosis level, HCV genotype and plasma biomarkers: Brain-Derived Neurotrophic Factor (BDNF), Interleukine 6 (IL6), Tumor Necrosis Factor (TNF-a),Glial fibrillary acidic protein (GFAP), Soluble CD14 (SCD14), Neuro-specific enolase (NSE).

The second neuropsychological assessment and clinical data collection is carried out after treatment, concretely 6 months after HCV is undetectable in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with indication to receive antiviral treatment
* Diagnosis of chronic infection by hepatitis C virus in the fibrous phase F3 or F4 that have not presented any clinical decompensation of their liver disease, with or without HIV co-infection

Exclusion Criteria:

* Active alcohol consumption> 40g daily or history of chronic alcoholism
* Active consumption of other toxics (heroin, cocaine, cannabis)
* Patients with minimum hepatic encephalopathy
* Background of cerebral neurological disease, chronic renal insufficiency and / or psychiatric illnesses assessed according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria, which can affect cognitive functions.
* Active use of psychotropics or benzodiazepines

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HCV patients who are candidates to direct antiviral treatment
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Memory tests | baseline, change at 6 months after treatment
  Rey Auditory Verbal Learning Test (RVLT, Spreen & Strauss 1998) assesses verbal learning, recall and recognition memory; Wechsler Adults Intelligence Scale III backward digits subtest (WAIS, Wechsler 1997) assesses working memory. All direct scores have been transformed into T-scores (mean=50; SD=10), which allows to obtain a single memory component.
Attention tests | baseline, change at 6 months after treatment
  Continous Performance Test (CPT, Conners 2000) assesses sustained attention, inattentiveness and impulsivity; WAIS forward digits subtest (WAIS III, Wechsler 1997) assesses attention. All direct scores have been transformed into T-scores (mean=50; SD=10), which allows to obtain a single attention component.
Executive function tests | baseline, change at 6 months after treatment
  Stroop Test (Stroop, 1935) assesses flexibility and inhibition of automatic responses; Trail Making Test (TMTA-B Reitan, 1993) assesses visual tracking and flexibility, phonetic and semantic fluency tests (Lezak, 1995) assess verbal fluency; Tower of London (Culbertson & Zillmer, 2005) assesses visual reasoning and planification. All direct scores have been transformed into T-scores (mean=50; SD=10), which allows to obtain a single executive function component.
Speed processing test | baseline, change at 6 months after treatment
  Digit symbol test (WAIS III, Wechsler 1997) assesses visuomotor speed. The direct scores have been transformed into T-scores (mean=50; SD=10).

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | baseline, change at 6 months after treatment
  It is a self-registering scale of 14 items: 7 items evaluating anxiety and 7 items evaluating depression (Zigmond & Snaith, 1983).
  Scoring range: 0-21 for each subscale. Scores >10 in each subscale imply a significant anxious/depressive symptomatology.
36-Item Short Form Health Survey (SF-36 ) | baseline, change at 6 months after treatment
  It is a self-registered scale for the assessment of quality of life ( Alonso y cols. , 1995). It consists on 8 dimensions: Physical functioning, limitations for physical issues, corporal pain, social functioning, mental health, limitations for emotional issues, vitality and general perception of the own health. For each dimension, the scoring range goes from 0 to 100, where higher values represent better outcome (better quality of life/less limitations/better functioning).
Fibroscan | Baseline, change at 6 months after treatment
  Degree of fibrosis: Speed of propagation of elastic waves measured with fibroscan.
HCV RNA | Baseline, change at 3 months after treatment, change at 6 months after treatment.
  Viral load quantity measured by plasma HCV RNA is collected in HIV co-infected patients
Immunosuppression state | Baseline
  The next cells were analyzed in blood, in HIV co-infected patients : CD4, %CD4, nadir CD4, CD8, % CD8, CD4/CD8 ratio.

OTHER OUTCOMES:
Blood Biomarkers measures | 1 day pretreatment and change at 6 months post treatment
  The next blood biomarkers were collected: Brain-derived neurotrophic factor (BDNF); Interleukine 6 (Il-6); Tumor Necrosis Factor (TNF-a ); Glial fibrillary acidic protein (GFAP); Soluble SCD 14 (sCD14) ; Neuro-specific enolase (NSE).